CLINICAL TRIAL: NCT05578430
Title: Neoadjuvant Immune-Checkpoint Blockade Therapy Combining With TACE For Resectable Hepatocellular Carcinoma With High Recurrence Risk: A Phase II, Single-arm Clinical Trial
Brief Title: AK104 Combining With TACE for Resectable Hepatocellular Carcinoma (MORNING)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC2022
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Resectable Hepatocellular Carcinoma
Keywords: Resectable Hepatocellular Carcinoma; Neoadjuvant Treatment; Immune-checkpoint Blockade; TACE
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE+Cadonilimab+Surgery (Experimental): After appropriate screening and randomization, patients enrolled will receive TACE plus 2-cycle of Cadonilimab treatment before surgery. Four weeks later after surgery, Cadonilimab treatment will be followed up to 16 cycles.
  Interventions: Drug: Cadonilimab; Procedure: TACE; Procedure: Surgery

INTERVENTIONS:
Drug: Cadonilimab — 10mg/kg by intravenous infusions every 3 weeks
  Other Names: AK104
Procedure: TACE — TACE will be performed per institutional standard of care.
Procedure: Surgery — Surgery will be performed per institutional standard of care.

SUMMARY:
This is a Phase 2, open-label, single-arm study of neoadjuvant immune-checkpoint blockade therapy (AK104) combining with TACE for resectable hepatocellular carcinoma. The purpose is to investigate the efficacy and safety of this therapeutic regimen to reduce the risk of postoperative recurrence in resectable HCC patients with a high risk of recurrence.

DETAILED DESCRIPTION:
The trial will recruit 54 patients. At the first step, 26 patients will be recruited. Only when at least 10 patients achieve major pathological response after surgery will the trial enter the second step and continue to recruit other patients. After being enrolled, all patients giving written informed consent will receive TACE plus 2-cycle of Cadonilimab treatment before surgery. Four weeks later after surgery, Cadonilimab treatment will be followed up to 16 cycles. The tumor response evaluation will be conducted on a regular basis until progression of disease. Long-term survival follow up will be conducted as well.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years but ≤75 years
2. Resectable HCC staged BCLC A/B
3. Treatment naïve for HCC
4. High risk for recurrence, meeting at least one of the following criteria:

   1. Multiple tumor lesions
   2. Individual tumor > 5cm
   3. AFP > 400 ug/L
   4. MVI positive based on preoperative MRI according to MVI predictive model of Radiomics
5. Measurable or evaluable lesions according to RECIST v1.1 criteria
6. ECOG performance status 0-1
7. Child-Pugh class A
8. Life expectancy ≥ 12 weeks
9. Adequate organ and marrow function as defined below:

   1. Hemoglobin ≥9.0 g/dL
   2. Absolute neutrophil count ≥ 1,500/μL
   3. Platelets count ≥ 75,000/μL
   4. Total serum bilirubin ≤ 1.5 ×upper limit of normal(ULN)
   5. AST and ALT ≤ 5 × ULN, ALP ≤ 4 ×ULN
   6. Serum creatinine ≤ 1.5 ×ULN
   7. INR ≤ 1.5 ×ULN, APTT ≤ 1.5 ×ULN
   8. Serum albumin ≥3.0 g/dL
10. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test.
11. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen as assessed by the treating investigator are eligible for this trial.
12. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Any prior treatment for HCC.
2. Tumor rupture or bleeding. Suspected abdominal metastasis.
3. A major surgical procedure, open biopsy, or significant traumatic injury with poorly healed wound within 6 weeks prior to enrollment.
4. History of allogenic organ transplantation.
5. Under other clinical trials.
6. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion: vitiligo or alopecia, hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement, any chronic skin condition that does not require systemic therapy or celiac disease controlled by diet alone.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to AK104 or other immune checkpoint inhibitors.
8. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection (including tuberculosis), uncontrolled hypertension (defined as blood pressure of > 140/90 mmHg during the screening period despite medical management), interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
9. History of hepatic encephalopathy, refractory ascites or esophagogastric varices with high risk of bleeding. Upper gastrointestinal hemorrhage within the year prior to the first dose of study drug.
10. Active hepatitis B infection without treatment (positive HBV surface antigen (HBsAg) and HBV DNA ≥ 1000 IU/ml). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Active hepatitis C infection (positive HCV antibody and HCV RNA above the lower limit of detection).
11. A primary brain tumor (excluding meningiomas and other benign lesions), any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, or history of a stroke within the year prior to the first dose of study drug.
12. History of active primary immunodeficiency.
13. History of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
14. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of study agent. The following are exceptions to this criterion: Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection). Systemic corticosteroids at physiologic doses that do not exceed 10 mg/day of prednisone or its equivalent. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
15. Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug. Note: Patients, if enrolled, should not receive live vaccine whilst receiving study drug and for at least 30 days after the last dose of study agent.
16. Systemic immunostimulant therapy within 14 days prior to the first dose of study agent.
17. History of serious systemic disease, including myocardial infarction or unstable angina within the 12 months prior to the first dose of study drug, hypertensive crisis or hypertensive encephalopathy, New York Heart Association (NYHA) grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication, significant vascular disease or symptomatic peripheral vascular disease.
18. History of coagulopathy, bleeding diathesis, or thrombosis within the 12 months prior to the first dose of study drug.
19. A serious, non-healing wound, ulcer, or bone fracture.
20. Pregnancy or lactation.
21. Total parenteral nutrition.
22. Exclusion from the study by the judgement of investigators, due to some factors that may lead to the forced termination of the study, including other acute, chronic or psychological disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response Rate (MPR rate) | Up to 2 years
  MPR rate is defined as the percentage of patients with over 90% of histological tumor tissue necrosis removed after neoadjuvant TACE combined with AK104 treatment.

SECONDARY OUTCOMES:
1-year recurrence rate | The percentage of patients who suffer recurrence one year after surgery.
  Up to 1 years
Objective response rate (ORR) | ORR is defined as the percentage of patients who have achieved complete response (CR) or partial response (PR), as measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, after neoadjuvant TACE combined with AK104 treatment but before
  Up to 2 years
Incidence of Adverse Events (AE) | The percentage of patients who suffer grade 3 or worse adverse events from the first dose of administration to last follow-up, assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
  Up to 2 years